CLINICAL TRIAL: NCT05812196
Title: Changes in the Respiratory System in Post-COVID Syndrome
Brief Title: Late Respiratory Consequences of SARS-CoV-2 Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Barna Babik, Professor, Szeged University
Other Study IDs: Post-COVID-Szeged
Record Dates: First submitted 2023-04-12; First posted 2023-04-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Function Tests; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID: Patients with COVID-19 infections.
  Interventions: Diagnostic Test: Lung function test; Biological: COVID infection
- Control: Patients without earlier diagnosis of COVID-19.
  Interventions: Diagnostic Test: Lung function test

INTERVENTIONS:
Diagnostic Test: Lung function test — Spirometry to assess lung volumes, forced oscillations to measure respiratory mechanics, whole body plethysmography to assess static lung volumes and airway resistance, lung diffusion capacity measurements.
Biological: COVID infection — Verified COVID-19 infection.
  Groups: Post-COVID

SUMMARY:
The goal of this observational study is to learn about the respiratory system in post-COVID syndrome. The main question aims to answer:

how the post-COVID syndrome alters the lung function Participants will be asked to perform lung function tests. Researchers will compare post-COVID group to matched control healthy individuals.

ELIGIBILITY:
Inclusion Criteria: COVID-19 infections in the post-COVID group. -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients after COVID-19 infection. In the control group, healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory mechanics | 6-12 months after COVID-19 infections
  Mechanical properties of the airways and respiratory tissues

SECONDARY OUTCOMES:
Spirometry | 6-12 months after COVID-19 infections
  Forced expiratory lung volumes
Lung diffusion capacity | 6-12 months after COVID-19 infections
  DLCO
Plethysmography | 6-12 months after COVID-19 infections
  Measurement of functional residual capacity and airway resistance by using a whole body plethysmograph.

CONTACTS AND LOCATIONS:
Locations (1):
- Barna Babik, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palfi A, Balogh AL, Polonyi G, Schulcz D, Zollei E, Bari G, Fodor GH, Barath K, Somfay A, Petak F, Babik B. Post-COVID changes in lung function 6 months after veno-venous extracorporeal membrane oxygenation: a prospective observational clinical trial. Front Med (Lausanne). 2023 Dec 20;10:1288679. doi: 10.3389/fmed.2023.1288679. eCollection 2023. PMID 38173937